CLINICAL TRIAL: NCT01523574
Title: Randomized, Placebo Controlled Study of Vitamin E for Oxaliplatin-induced Neuropathy Prophylaxis
Brief Title: Vitamin E for Oxaliplatin-induced Peripheral Neuropathy Prophylaxis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Felipe Melo Cruz (Other)
Responsible Party: Sponsor-Investigator, Felipe Melo Cruz, Director, Faculdade de Medicina do ABC
Organization: Faculdade de Medicina do ABC (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VE01
Record Dates: First submitted 2011-12-19; First posted 2012-02-01 (Estimated); Last update posted 2012-02-01 (Estimated); Status verified 2012-01

CONDITIONS: Peripheral Neuropathy
Keywords: oxaliplatin; vitamin e; neuropathy; peripheral; prophylaxis
MeSH Terms: conditions — Peripheral Nervous System Diseases | interventions — Vitamin E; Calcium Gluconate; Lead; Magnesium Sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Group (Placebo Comparator): Five days before chemotherapy:1 x daily Used until one week after third oxaliplatin infusion: 1 x daily
  Interventions: Drug: Placebo
- Vitamin e (Experimental): Five days before chemotherapy:1 x daily Used until one week after third oxaliplatin infusion: 1 x daily
  Interventions: Drug: Vitamin E

INTERVENTIONS:
Drug: Vitamin E — Vitamin E 400mg PO orally
  Other Names: Calcium gluconate 1g, IV, before and after oxaliplatin; Magnesium sulfate 1g, IV, before and after oxaliplatin
  Arms: Vitamin e
Drug: Placebo — Placebo, given orally
  Other Names: Calcium gluconate 1g, IV, before and after oxaliplatin; Magnesium sulfate 1g, IV, before and after oxaliplatin
  Arms: Control Group

SUMMARY:
Introduction: Oxaliplatin (Ox) is a frequently used platinum-based medication that is a part of many chemotherapy regimens for the treatment of several gastrointestinal malignancies. One of the most important limitations to its use is the induction of both acute and chronic peripheral neuropathy (PN). Previous studies have shown that vitamin E can reduce the incidence of cisplatin-induced PN by 50%. In this study, the investigators aimed to determine if vitamin E could also prevent Ox-induced acute PN

DETAILED DESCRIPTION:
This was a prospective, phase II, randomized pilot study. Patients were randomized 5 days before the start of Ox to receive either vitamin E at 400 mg daily or placebo, until after the end of the Ox-based chemotherapy regimen. The investigators evaluated PN intensity using the CTCAE version 3 and specific Ox PN gradation scales. The investigators included patients with colorectal and gastric cancers scheduled to receive Ox-based chemotherapy. Both groups received calcium and magnesium supplements before and after oxaliplatin infusions.

ELIGIBILITY:
Inclusion Criteria:

* ECOG Performance status 0 or 1
* Older than 18 years
* New diagnose with colorectal or gastric cancer
* Scheduled to receive oxaliplatin-based regimens

Exclusion Criteria:

* Excluded patients with a previous history of PN or with symptomatic PN at entry into the study
* Excluded patients who received other chemotherapy regimens (except isolated 5-fluorouracil)
* Patients currently receiving gabapentin, carbamazepine, amitriptyline, amifostine or multivitamins

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2009-08; Primary Completion 2010-11 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Incidence and grade of Peripheral neuropathy by common terminology criteria for adverse events v 3.0(CTCAE)and specific Ox PN gradation scales. | Within the first 45 days (plus or minus 7 days) of treatment ( 3 x oxaliplatin infusions)

CONTACTS AND LOCATIONS:
Overall Officials: Auro del Giglio, phD, Study Director — Faculdade de Medicina do ABC
Locations (1):
- Faculdade de Medicina do ABC, Santo André, São Paulo, Brazil

REFERENCES:
- [Derived] Afonseca SO, Cruz FM, Cubero Dde I, Lera AT, Schindler F, Okawara M, Souza LF, Rodrigues NP, Giglio Ad. Vitamin E for prevention of oxaliplatin-induced peripheral neuropathy: a pilot randomized clinical trial. Sao Paulo Med J. 2013;131(1):35-8. doi: 10.1590/s1516-31802013000100006. PMID 23538593